CLINICAL TRIAL: NCT04165447
Title: Randomized Trial Evaluating the Effectiveness of Within Versus Across-Category Front-of-Package Lower-Calorie Labelling on Food Demand
Brief Title: Evaluating the Effectiveness of Within Versus Across-Category Front-of-Package Lower-Calorie Labelling on Food Demand
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke-NUS Graduate Medical School (Other)
Collaborators: National University of Singapore (Other)
Responsible Party: Principal Investigator, Eric A. Finkelstein, Principal Investigator, Professor, Duke-NUS Graduate Medical School
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Health Services Research
Other Study IDs: AG-2014-001
Record Dates: First submitted 2019-11-11; First posted 2019-11-18 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Food Selection
Keywords: nutrition; front-of-pack label; calories; online grocery store; diet; groceries; obesity
MeSH Terms: conditions — Food Preferences; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No labeling Control (No Intervention): Arm 1 was the Control condition, which did not display the label on any products.
- Within-category labeling (Experimental): Arm 2 displayed the label on the 20% of products that were lowest in calories per serving within each product category (termed Within-category Labeling, WC).
  Interventions: Behavioral: Front-of-pack labeling strategy
- Across-category labeling (Experimental): Arm 3 displayed the label on the 20% of all products that were lowest in calories per serving (termed Across-category Labeling, AC).
  Interventions: Behavioral: Front-of-pack labeling strategy

INTERVENTIONS:
Behavioral: Front-of-pack labeling strategy — We designed a simple 'Lower Calorie' directive logo. We labeled the 20% of products with the lowest calories per serving within or across categories. All serving sizes used in this study were the average of the serving sizes within each category. Prior to conducting the analysis, we standardized the serving size by using the mean serving size within each subcategory. This standardization ensures that similar products are compared equally as serving sizes can be arbitrarily set by the manufacturers. The labels were displayed below the product images.
  Arms: Across-category labeling; Within-category labeling

SUMMARY:
The important role that diet plays in health and disease is well established, as is its association with rising rates of obesity-a phenomenon of increasing concern in Singapore. Changes in lifestyle patterns, including a movement towards a more western-style diet with an emphasis on pre-packaged and fast food, have contributed to the upward trend in weight. This study aims to test two competing approaches for calorie labelling in efforts to reduce total calories purchased. In Arm 1 (termed across category labelling) a low calorie logo will be displayed on the 20% of products on the web store that are lowest in calories per serving. Arm 2 will display this logo on the 20% of products that are lowest in calories per serving within each product category (termed within category labelling). Arm 3 is the Control condition which will not display any logo on any products.

For our primary outcome, the investigators hypothesize that the proportion of labelled products (or those that would have been labelled if not in control arm) purchased in each intervention arm will be greater than in control.

For secondary hypotheses the investigators expect the following ordering across the three (Control, Within category, Across category) arms:

1. total calories (adjusted for household size): C > A > W
2. calories per serving: C > A > W
3. calories per dollar spent: W > A > C
4. total dollars spent (adjusted for household size) : W > A > C

DETAILED DESCRIPTION:
For this study an online grocery store was developed that contains over 3200 products commonly purchased in local supermarkets. The products available for purchase include foods from many different categories such as dairy products, snacks, processed meats and soft drinks. The web-based grocery store was designed to mirror an actual web-based grocery store in look and feel. All products include a picture of the item, current retail price, the Lower Calorie logo (where applicable), and other package size and nutrition information currently required for products in Singapore. The online grocery store features a grocery cart that shows the items purchased. The NUS Online Collection Facility payment system has been integrated with the online grocery store for participants to make payments.

Study design: This will be a crossover study design with all participants exposed once to 3 shopping conditions (1xControl, 1xIntervention 1 (I1), 1x Intervention 2(I2)) in random order. The total study duration for each participant is 3 weeks, with each participant spending 1 week in each shopping condition.

For the Control condition the participants are not exposed to the lower calorie logo. For Intervention 1 (Across), the participant will see the lower calorie logo applied to foods with the lowest calories per serving across all food categories. For intervention 2, the participant will see the lower calorie logo applied to the 20% of foods with the lowest calories per serving within each food category. These foods will be tagged with the 'Lower Calorie' logo.

Participants will be asked to shop once a week during each of the 3 weeks of the study, and will therefore shop for a total of 3 times during the study. This will include 1 shop within each shopping condition (control, I1, and I2). Participants will purchase and receive at least 1 and up to 3 of their grocery orders. This ensures that purchases will be an accurate reflection of their actual shopping experience.

Since there are 3 shopping conditions (Control, I1, and I2) and the specific weeks that the participant's shopping trips will be pre-determined for purchase (but unknown to participants), each participant will be randomly assigned at baseline to 1 of 6 groups that vary the sequence of shopping conditions and which shops will result in an actual food delivery.

For each shop there will be a minimum spend of SGD50 and a maximum spend of SGD250. A minimum spend ensures that participants complete a typical weekly grocery order. A maximum spend is to make the study more manageable given foods will need to be reordered and delivered. The grocery orders that participants purchase will be ordered by Duke-NUS using RedMart, a popular online grocery store in Singapore, and RedMart will deliver the grocery items. The store was created using products currently available on the RedMart website to allow us to repurchase from a single location.

Redmart is engaged in this project as our collaborator. As such, the relationship between the Parties is that of independent contractor and contractee. Neither party is an agent of the other nor have any right or authority to create any obligation or responsibility on behalf of the other. Neither is Duke-NUS in any way endorsing or marketing the services of Redmart.

At the end of the study participants who have completed all 3 shops as instructed will receive a RedMart e-Voucher worth $75 payment that can be redeemed against any products on RedMart.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 21 years and above
* Primary grocery shopper for the household
* Registered RedMart (an online grocery store) shoppers

Exclusion Criteria:

* Under 21 years of age
* Not the primary grocery shopper for the household
* Not a resident in Singapore
* Not a registered online shopper of RedMart

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Proportion of the basket represented by Lower Calorie products per shopping trip | Once a week for three weeks
  Proportion of products that are designated as labelled in the interventions

SECONDARY OUTCOMES:
Calories purchased per dollar spent per shopping trip | Once a week for three weeks
  Calories purchased per dollar spent in kcal per $
Total spending per shopping trip | Once a week for three weeks
  Total spending ($)
Total calories purchased per shopping trip | Once a week for three weeks
  Total calories purchased (in kcal)
Calories per serving per shopping trip | Once a week for three weeks
  Calories per serving (in kcal/serving)

CONTACTS AND LOCATIONS:
Locations (1):
- Duke-NUS Medical School, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
The datasets used and/or analysed during the current study are available from the corresponding author on reasonable request. All data will be de-identified.
Supporting Information: Study Protocol, ICF, CSR, Analytic Code
Time Frame: Up to 10 years after study conclusion.
Access Criteria: Reasonable request.

REFERENCES:
- [Derived] Finkelstein EA, Ang FJL, Doble B. Randomized trial evaluating the effectiveness of within versus across-category front-of-package lower-calorie labelling on food demand. BMC Public Health. 2020 Mar 12;20(1):312. doi: 10.1186/s12889-020-8434-1. PMID 32164634